CLINICAL TRIAL: NCT01274364
Title: China-JD Program: A Multi-centre Demonstration Project to Evaluate the Effectiveness and Acceptability of the Joint Asia Diabetes Evaluation (JADE) and DIAbetes MONitoring Database (DIAMOND) Programs in Asian Type 2 Diabetic Patients
Brief Title: Establishing a Diabetes Registry Using the JADE-DIAMOND Electronic Portal (CN001)
Acronym: China-JD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asia Diabetes Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRE-2010-112
Record Dates: First submitted 2011-01-09; First posted 2011-01-11 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Diabetes
Keywords: Diabetes; Structured Care
MeSH Terms: conditions — Diabetes Mellitus | interventions — Diamond

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- JADE (Experimental): Patients will receive comprehensive assessments at baseline and again after 12-months. In the interim between these two time points patients will receive protocol-driven diabetes care using a web-based disease management program (JADE), delivered by a trio-team comprising of a trained doctor, nurse and physician assistant.
  Interventions: Other: JADE
- DIAMOND (Active Comparator): Patients will receive comprehensive assessments at baseline and again after 12-months. In the interim between these two time points patients will be managed according to 'usual care' procedures.
  Interventions: Other: DIAMOND

INTERVENTIONS:
Other: JADE — Patients will receive comprehensive assessments at baseline and again after 12-months. In the interim between these two time points patients will receive protocol-driven diabetes care using a web-based disease management program (JADE), delivered by a trio-team comprising of a trained doctor, nurse and physician assistant.
  Arms: JADE
Other: DIAMOND — Patients will receive comprehensive assessments at baseline and again after 12-months. In the interim between these two time points patients will be managed according to 'usual care' procedures.
  Arms: DIAMOND

SUMMARY:
Quality diabetes care requires a team approach and informed decisions of patients and care providers. Several lines of evidence suggests that a protocol-driven care model delivered by trained staff with focus on periodic assessments, reinforcement of patient compliance and attainment of multiple treatment targets reduces risk of cardio-renal complications and early death in type 2 diabetes.

The investigators hypothesize that the use of state of the art information technology to record, manage and analyze the large amount of clinical information generated during various consultation visits will improve the effectiveness and efficiency in implementing these care protocols through decision support and regular feedback to both patients and care team.

DETAILED DESCRIPTION:
Diabetes is now a pandemic disease affecting 5-10% of global population. More than 60% of affected people will come from Asia with the number expected to increase from 85 million in 2005 to 132 million in 2010 in Asia alone. On average, diabetes reduces life expectancy by 10-12 years. While stroke, heart disease and kidney failure account for more than 50% of global deaths, 30-50% of patients with these conditions have diabetes as a major contributing factor. In contrast to the West, the main increase in diabetes prevalence in Asia will occur in the young to middle aged population. On average, 17 million people die from stroke and heart disease on a yearly basis. Of these, 11 million occur in Asia, affecting many young parents and economically active people.

Despite their devastating nature, many diabetic complications can be prevented and managed effectively to preserve health, reduce disabilities and improve quality of life. However, there are multiple barriers in the implementation of quality diabetes care. These include insufficient knowledge base of health care professionals, fragmented nature of health care systems, lack of reimbursement for outpatient procedures including therapeutic patient education, poor compliance to treatment in part due to the silent nature of diabetes and associated complications as well as the complex nature of care protocols. The latter include periodic evaluation of clinical and laboratory parameters and the need for people with diabetes to adhere to long term medications and self care.

While optimal management of risk factors and treatment to targets can substantially reduce the risk of diabetes associated complications, the challenge lies in the effective translation of this evidence to clinical practice. Since mid 1990s, inspired by the benefits of structured care, made possible during the conduct of clinical trials, the CUHK Diabetes Care & Research Group has developed prototypes of structured care protocols including an annual comprehensive assessment using a doctor-nurse-physician assistant team. Consistent with international data, these prototypes substantially improve rates of treatment compliance and attainment of multiple treatment targets resulting in reduced death and cardio-renal complication rates.

The Joint Asia Diabetes Evaluation (JADE) Program is a web-based disease management program conceptualized, developed and tested by the Asia Diabetes Foundation (ADF) since 2007, supported by a MSD educational grant. The objectives of the JADE Program include:

1. to promote collective learning and sharing of best practices in diabetes based on regionally relevant evidence
2. to increase regional awareness about the magnitude of diabetes and its preventable nature through education, ongoing data collection and implementation of evidence-based guidelines
3. to establish a regional diabetes registry
4. to collect the evidence base to inform relevant stakeholders including public, people with diabetes, health care professionals, policy makers and payors to change policies and practices in order to make quality diabetes care accessible, sustainable and affordable.

Using state of the art information technology, the JADE and DIAMOND electronic portal provides a virtual platform to enable care professionals to record, manage and analyse the large amount of information collected during various consultation visits. The Programs also incorporate risk equations developed and validated by the CUHK Diabetes Care & Research Group to help doctors assess their patients' future event rates. This information, displayed in charts and trend lines, can be communicated to patients and doctors to motivate behavioral changes and encourage dialogues to set treatment goals.

Apart from providing templates for documentation of risk factors and complications using standardized protocols, the JADE Program also incorporates different evidence-based care protocols with recommendations on follow up schedules and care processes in accordance to the patient's risk profile. Decision support in terms of prompts, charts, trend lines and practice tips are used to help doctors and patients to make informed decisions and to optimize care. The JADE Program also possesses matrixes which enable care providers to track clinical progress and risk factor control for benchmarking and quality improvement purposes. On the other hand, the DIAMOND Program provides the first step to entry of a quality assurance program by establishing a diabetes registry at a clinic level. The ongoing collection of these data provides an invaluable platform for collaborative epidemiological and interventional studies pertinent to Asian populations.

In this multicentre study, we shall use a trio team consisting of a trained doctor, nurse and physician assistant (PA) to deliver protocol-driven diabetes care using a web-based disease management program, the Joint Asia Diabetes Evaluation (JADE) Program. To fully realize the functionality of the JADE Program requires changes in the practice environment and deployment of additional manpower (e.g. a nurse and a PA) to enter data and provide reminders to patients and doctors to improve adherence to protocols. In settings where these changes may not be immediately possible, periodic comprehensive assessment using the structured template in the JADE Program allows recognition of risk factors and complications for early intervention. The latter will allow data collected in a systematic manner which forms the basis of a DIAbetes MONitoring Database (DIAMOND) as a first step towards quality assurance.

After explanation by trained doctors and nurses and with written informed consent, patients will be randomized to either the JADE or DIAMOND Program. The former encompasses all components of the structured care delivered by a trio-team of doctor, nurse and PA while the DIAMOND Program only consists of comprehensive assessments at baseline and 12-month with patients managed in the usual manner thereafter. At the end of 12 months, all patients will undergo repeat comprehensive assessments for comparison of rates of attainment of treatment targets, behavioral changes, quality of life and default rates.

Aims of the study:

1. To evaluate the reach, adoption and acceptability of the JD Program by patients and health care team;
2. To compare the effectiveness of the JADE (structured care) versus DIAMOND (usual care) Programs in attainment of treatment targets, improvement of quality of life and changes in behaviors;
3. To document the pattern of complications, risk factors, use of medications and quality of life in type 2 diabetic patients

Study sites:

1. Beijing People's Hospital, Beijing
2. Peking Union Hospital, Beijing
3. 1st Hospital, Peking University Hospital, Beijing
4. China-Japan Friendship Hospital, Beijing
5. Shanghai Sixth People's Hospital, Shanghai
6. Third Affiliated Hospital of Sun Yat-Sen University, Guangzhou

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic patients attending hospitals or affiliated clinics led by PIs of the JADE Program who are living in the area with an intention to have 'regular' follow-up
* Aged >18 years
* Patients can have newly diagnosed or established disease, treated with lifestyle or blood glucose lowering drugs including oral agents with or without insulin
* For newly diagnosed type 2 diabetic patients, their plasma glucose levels should be: a) Fasting plasma glucose (PG) >7.0 mmol/L on 2 or more occasions, and/or b) Random (or post-OGTT 2h) PG >11.1 mmol/L on 2 or more occasions, and/or c) HbA1c >6.5%

Exclusion Criteria:

* Type 1 diabetes defined as a history of ketosis at diagnosis [acute symptoms with heavy ketonuria (>3+) or ketoacidosis] or continuous requirement of insulin within one year of diagnosis
* Patients with reduced life expectancy (e.g. less than 6-months) due to recent diagnosis of advanced cancers (e.g. within last 2 years) and other life threatening conditions
* Patients with a mental condition rendering them unable to understand the nature, scope, and possible consequences of the study
* Patients actively enrolled in another intervention study
* Patients who are unwilling to return for regular follow up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3586 (Actual)
Dates: Start 2010-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who attain 2 or more of the 'ABC' targets | 12 months
  Percentage of patients who attain 2 or more of the following 3 targets:
  * HbA1c <7%
  * BP <130/80 mmHg
  * LDL cholesterol <2.6 mmol/L

SECONDARY OUTCOMES:
New onset of all diabetes-related endpoints | 12 months
  This includes;
  * cardiovascular endpoints (acute myocardial infarction, revascularisation procedures, heart failure or unstable angina or arrhythmia requiring hospital admissions, lower extremity amputation or foot ulcers)
  * chronic kidney disease (eGFR<60 ml/min/1.73m2) and end stage renal disease (dialysis and/or eGFR<30 ; ml/min/1.73m2)
  * visual impairment (corrected visual acuity of 20/200 or lower) or eye surgery;
  * cancer
  * any hospitalization due to complications related to diabetes and/or its treatment (such as hypoglycaemic attacks)
  * death
Quality of Life | 12 months
Frequency of hypoglycaemia (in the last 3 months) | 12 months
Behavioral changes (in the last 3 months) | 12 months
  1. Frequency of Self Blood Glucose Monitoring
  2. Adherence to balanced eating
  3. Adherence to regular exercise
  4. Adherence to recommended procedures (e.g. return for blood tests or education classes)
Number of hospitalizations, follow up visits by doctors and other care professionals | 12 months
Default rates at end of study | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Juliana Chan, MD, Principal Investigator — Asia Diabetes Foundation
Locations (1):
- Asia Diabates Foundation, Shatin, Hong Kong

REFERENCES:
- [Derived] Tutino GE, Yang WY, Li X, Li WH, Zhang YY, Guo XH, Luk AO, Yeung RO, Yin JM, Ozaki R, So WY, Ma RC, Ji LN, Kong AP, Weng JP, Ko GT, Jia WP, Chan JC; China JADE Study Group. A multicentre demonstration project to evaluate the effectiveness and acceptability of the web-based Joint Asia Diabetes Evaluation (JADE) programme with or without nurse support in Chinese patients with Type 2 diabetes. Diabet Med. 2017 Mar;34(3):440-450. doi: 10.1111/dme.13164. Epub 2016 Jul 11. PMID 27278933
- See also: Works of the Asia Diabetes Foundation, including the DIAMOND program. — http://www.adf.org.hk